CLINICAL TRIAL: NCT03044834
Title: Review of the Paediatric Pleuropulmonary Blastoma French Series
Acronym: PPB
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC15_3009_PPB; 15.18 (Other: Comité d'Ethique Régional de Rennes); 15.468 (Other: CCTIRS); 915465 (Other: CNIL)
Record Dates: First submitted 2017-01-16; First posted 2017-02-07 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Pleuropulmonary Blastoma
MeSH Terms: conditions — Pleuropulmonary blastoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pleuropulmonary Blastoma: * Patients born between 01/01/2000 and 01/01/2016 ;
  * Followed up for PPB
  * Treated in a French department of paediatric oncology or paediatric surgery
  * Study agreement
  Interventions: Other: PPB

INTERVENTIONS:
Other: PPB — Global current care

SUMMARY:
Pleuropulmonary blastoma is a rare embryonic malignant tumour that remains the most frequent malignant tumour of the lung in childhood. The International Pleuro pulmonary Blastoma Registry (IPPB) found only 220 cases in 2009 and 350 in 2015. In France, 20 cases were identified in 2009.

Three histologies are described: type 1 purely cystic, type 2 combined and type 3 solid. Median age at diagnostic is 12 months, 35 months and 41 months respectively. Evolution is possible from type 1 to type 2 or 3 in 10% of the cases.

Since 2009, DICER 1 mutations research is proposed systematically to all families.

PPB symptoms are usually non-specific. Diagnostic is evoked when imaging work up shows bubbles or solid lesions, and confirmed by pathological analysis. However the diagnosis can be difficult because of the proximity with congenital cystic adenomatoid malformation.

The French society of paediatric oncology recommends surgery at first instance. PPB type 1 remains a problem because some are still misdiagnosed as CCAM, a benign lesion. Chemotherapy depends on the PPB type and the quality of the resection. There is a real interest to analyse the French series.

The prognosis of type 2 and 3 is low with a 5 years survival rate of 45-60%, whereas type 1 survival rate is 91%. The French experience reports a 100% survival rate in type 1 and 48% in type 2 and 3. Other prognostic factors are initial size of the tumour, extra pulmonary invasion and quality of surgery.

Early local relapses are possible and late ones concern more often type 2 and 3 with more cerebral metastasis.

In 2009, the french cases were collected, but no update has been performed since. The aim of this retrospective review of the cases since 2000, is to audit the care of PPB patients in France and update the French rare tumour database.

Evoking PPB diagnosis is difficult when imaging shows a neonatal cystic lesion. There are no radiologic criteria in the literature that differentiate congenital pulmonary cystic lesion and PPB type 1. Radiological presentation is however overlapping. Another aim of this study will be to look for a predictive sign of type 1 PPB.

DETAILED DESCRIPTION:
Multicentre retrospective study

ELIGIBILITY:
Inclusion Criteria:

* Patients born between 01/01/2000 and 01/01/2016 ;
* Followed up for PPB
* Treated in a French department of paediatric oncology or paediatric surgery
* Study agreement

Exclusion Criteria:

* Part of the care out of France
* Study disagreement

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients born between 01/01/2000 and 01/01/2016, followed up for PPB, treated in a French department of paediatric oncology or paediatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2018-02-22 (Actual); Study Completion 2018-07-09 (Actual)

PRIMARY OUTCOMES:
Overall survival | Within 5 years from the diagnosis
Progression free survival | Within 5 years from the diagnosis
  Characterize the evolution and the global care of PPB in the French series

SECONDARY OUTCOMES:
State of PPB surgical care | Within 5 years from the diagnosis
Radiology sign | Within 5 years from the diagnosis
  Identification of a type 1 PPB predictive radiological sign

CONTACTS AND LOCATIONS:
Overall Officials: Alexis ARNAUD, MD, Principal Investigator — Rennes University Hospital
Locations (18):
- France (18):
  - Angers University Hospital, Angers
  - Bordeaux University Hospital, Bordeaux
  - Caen University Hospital, Caen
  - Grenoble University Hospital, Grenoble
  - Kremlin-Bicêtre Hospital, Le Kremlin-Bicêtre
  - Lille University Hospital, Lille
  - Lyon Universty Hospital, Lyon
  - Marseille University Hospital, Marseille
  - Montpellier University Hospital, Montpellier
  - Nantes University Hospital, Nantes
  - Nice University Hospital, Nice
  - Necher Hospital, Paris
  - Poitiers University Hospital, Poitiers
  - Curie Institute, Saint-Cloud
  - Réunion University Hospital, Saint-Paul
  - Toulouse University Hospital, Toulouse
  - Tours University Hospital, Tours
  - Gustave Roussy Institute, Villejuif